CLINICAL TRIAL: NCT06309810
Title: Stereotactic Radiosurgery (SRS) in Malignant Spasticity and Hypertonia: a Pilot Study
Brief Title: Stereotactic Radiosurgery (SRS) in Malignant Spasticity and Hypertonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-35
Record Dates: First submitted 2023-06-20; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Spasticity/Paresis
MeSH Terms: conditions — Muscle Spasticity; Paresis | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Experimental): The treatment will be administered with a TrueBeam™ (Varian Medical Systems, Palo Alto, CA, USA) linac, equipped with a Millenium 120-leaves MLC.
  The target will be represented by 5 mm of the specific spinal nerve responsible for the spams. A lateral 1 mm margin will be added to the target to generate the corresponding planning treatment volume (PTV). The prescribed dose will be 45-60 Gy in a single fraction. The treatment dose will be chosen based on patients' general condition, and possibility to respect the dose limits (constraints) for the organs at risk (OARs).
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — The treatment will be administered with a TrueBeam™ (Varian Medical Systems, Palo Alto, CA, USA) linac, equipped with a Millenium 120-leaves MLC.
  The target will be represented by 5 mm of the specific spinal nerve responsible for the spams. A lateral
  1 mm margin will be added to the target to generate the corresponding planning treatment volume (PTV). The prescribed dose will be 45-60 Gy in a single fraction. The treatment dose will be chosen based on patients' general condition, and possibility to respect the dose limits (constraints) for the organs at risk (OARs).

SUMMARY:
This is a pilot, experimental, monocentric study. The main objective of the study is to evaluate whether stereotactic radiotherapy is able to reduce symptomatic spasticity from a clinical point of view, and therefore induce an improvement in posture and quality of life in patients with malignant spasticity.

The study foresees the enrollment of about 10 patients, in a period of 24 months. The radiotherapy treatment will be delivered in a single session with an image-guided stereotaxic technique, and a prescription dose between 45 and 60 Gy; subsequently the patients will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

* Malignant spasticity measured with the Modified Ashworth Scale (MAS≥3) or highly impairing spasticity and hypertonia (Numeric Rating Scale >8 scored by patient or care-giver)
* Age ≥ 18 years old
* Availability of a diagnostic MR scan of the spine segment of interest and electromyography of inferior limbs within 3 months prior to study entry
* Previous ineffective conventional treatment for spasticity or absence of others therapeutic strategies (i.e. negative baclofen pump test, comorbidity limiting the pump implant as spondylodiscitis or severe obesity)
* Plegic patients or minimally conscious state patient
* Signed informed consent (in case of minimally conscious state patients, consent form will be signed by her / his legal representative)

Exclusion Criteria:

* Age < 18 years old
* Previous radiation in the same anatomical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
MAS | 1 year after treatment
  Reduction of Modified Ashworth Scale (MAS) after SRS. A reduction of at least 1 point is considered for response evaluation.

SECONDARY OUTCOMES:
Acute and late toxicity (CTCAE) | 90 days from the RT treatment
  Acute and late toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE version 5.0). More specifically, acute toxicity will be defined as any event occurred within 90 days from the RT treatment while late toxicity will be defined as any event recorded after this time.
Quality of life (SF-12) | 1 year after treatment
  SF-12® Questionnaire will be administered to evaluate quality of life previously and after treatment (not applicable for patients in minimally conscious state).
Quality of nursing (VAS) | 1 year after treatment
  Visual Analogic Scale (VAS will be administered to the care-giver in minimally conscious state patient (VAS 1: many difficulties in nursing, VAS 10: none difficulties in nursing) before and after treatment.
Radiological characteristics and treatment-related changes of the spinal roots | 6 months after SRS
  The radiological characteristics and treatment-related changes of the spinal roots will be evaluated with multiparametric MR. Specific quantitative analyzed parameter will be: fractional anisotropy and diffusivity. Changes in morphology will be evaluated with a MR scan acquired 6 months after SRS.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria di Negrar, Negrar, Verona, Italy